CLINICAL TRIAL: NCT00196963
Title: Assess the Immunogenicity, Safety, Reactogenicity of 1 Dose of 4 Different Formulations of GSK Biologicals' Meningococcal Conjugate Vaccine (MenACWY) vs 1 Dose of Mencevax™ ACWY in Healthy Subjects Aged 15-19 Yrs
Brief Title: Evaluate 4 Different Formulations of Meningococcal Serogroups A, C, W-135, Y Conjugate Vaccine When Given as 1 Dose to Healthy Subjects Aged 15-19 Yrs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 103532
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Meningococcal
MeSH Terms: conditions — Meningococcal Infections | interventions — Meningococcal Vaccines

INTERVENTIONS:
Biological: Meningococcal (vaccine)

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, safety and reactogenicity of one dose of four different formulations of the MenACWY conjugate vaccine when given to healthy subjects aged 15-19 years. The selection of the best formulation will be based on data obtained up to one month after the vaccine dose.

DETAILED DESCRIPTION:
3 formulations of GSK's MenACWY conjugate vaccine will be administered in a double-blind manner, while the 4th one will be single-blinded. Administration of the candidate vaccine or of the active control (Mencevax™ ACWY) will be done in an open manner. Subjects will receive one vaccine dose (GSK's MenACWY conjugate vaccine or Mencevax™ ACWY vaccine), and will have 2 blood samples taken, before and one month after vaccination.

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female between, and including, 15 and 19 years of age at the time of vaccination.
* Written informed consent obtained. Subject with previously completed routine childhood vaccinations to the best of his/her knowledge or his/her parents'/guardians' knowledge.
* Female subjects should be of non-childbearing potential, or abstinent, or using an adequate contraception.

Exclusion criteria:

* Previous vaccination against OR history of OR exposure within previous 12 months to meningococcal serogroup A, C, W-135 or Y disease.
* Administration of a tetanus vaccine within 6 months before study vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of any neurologic disorders or seizures.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2005-03; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
% of serum bactericidal activity SBA-MenA, SBA-MenC, SBA-MenW-135 and SBA-MenY responders (i.e.>= 4-fold increase in SBA titre from pre to post vaccination) at 1 month after the vaccine dose.

SECONDARY OUTCOMES:
Prophylaxis meningococcal serogroups A, C, W-135, Y disease

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Thuin, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 103532 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103532 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103532 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103532 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103532 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register